CLINICAL TRIAL: NCT02010671
Title: Understanding a Woman's Choice of Mode of Delivery Before Initial Consult With Her Obstetrician After Having One Prior Cesarean Section
Brief Title: Survey of Women's Choice of Delivery Before Consulting With Her Obstetrician
Status: Terminated | Type: Observational
Why Stopped: Inadequate enrollment
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 477211
Record Dates: First submitted 2013-09-27; First posted 2013-12-13 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Pregnancy; Previous Cesarean Section
Keywords: Pregnancy; Cesarean Section; Survey; Delivery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with a prior cesarean section: Survey of women who had a cesarean section with their last pregnancy and no other prior cesarean section deliveries
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
We are surveying women who have had a previous cesarean section at the time of entry into prenatal care for their next pregnancy about their thoughts related to a trial of labor after cesarean (TOLAC) or repeat c-section.

DETAILED DESCRIPTION:
This is a survey for women who have had a previous cesarean section, also known as a c-section, with their last pregnancy. The study is looking at what factors and people may influence the decisions women make about their birthing plan after they have had a previous c-section. If they qualify, women will be asked to complete a brief survey at their initial Ob/Gyn appointment before they see their Ob doctor. In order to qualify, women must:

* Be pregnant
* Have not seen an obstetrician for this pregnancy
* Be at least 18 years old
* Be able to read English
* Have had a prior pregnancy delivered by c-section
* Only had one prior c-section
* The c-section must have been the last pregnancy before this one

Questions that will be asked include:

* Demographic information (examples: age, race/ethnicity)
* Pregnancy information
* Delivery questions
* Factors that may influence her birthing plan

Participants will also be asked if the study staff can follow up after her delivery to see what kind of delivery she had (vaginal or c-section).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women
* 18 years old or older
* Prior pregnancy with cesarean delivery
* No prior obstetric physician care during current pregnancy

Exclusion Criteria:

* More than one prior cesarean
* Women who cannot read English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the new obstetrics patients in the University of California, Davis Department of Obstetrics and Gynecology department clinics.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Participant Opinions of mode of delivery as compared to actual mode of delivery | Mode of delivery will be assessed after delivery, average 40 weeks gestational age (7-9 months after enrollment)
  Mode of delivery

SECONDARY OUTCOMES:
Factors that influence participant's opinion of mode of delivery | Collected at time of study enrollment, typically 4-12 weeks into the subject's pregnancy.
  Participants will be asked what influences their opinions of mode of delivery, such as significant other, clinicians, family, friends, or others. They will also be asked how much these factors may influence their decisions (high influence, some influence, no influence).

OTHER OUTCOMES:
Trust of information they receive | Collected at study enrollment, typically 4-12 weeks into the subject's pregnancy.
  Participants will be asked if they trust the information that they receive from influencing factors, such as significant others, clinicians, family, friends, or other.

CONTACTS AND LOCATIONS:
Overall Officials: Maricela Rangel-Garcia, Principal Investigator — University of California, Davis; Mitchell Creinin, MD, Study Director — University of California, Davis
Locations (1):
- University of California, Davis Department of Obstetrics and Gynecology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No